CLINICAL TRIAL: NCT01643681
Title: Safety and Efficacy of Autologous Adipose Tissue Derived Mesenchymal Stem Cells Transplantation in Patient With Lumbar Intervertebral Disc Degeneration
Brief Title: Autologous Adipose Tissue Derived Mesenchymal Stem Cells Transplantation in Patient With Lumbar Intervertebral Disc Degeneration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer willing to continue clinical trials
Sponsor: R-Bio (Industry)
Collaborators: Korea University Anam Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSC-MSCs-LIDD
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Lumbar Intervertebral Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AdMSC (Experimental): Autologous Adipose Tissue derived Mesenchymal Stem Cells
  Interventions: Procedure: Autologous Adipose Tissue derived MSCs Transplantation

INTERVENTIONS:
Procedure: Autologous Adipose Tissue derived MSCs Transplantation — Into lumbar intervertebral disc infusion of Autologous Adipose Derived Mesenchymal Stem Cells. Dose : 4x10e7 cells/1mL

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous transplantation of Adipose Tissue derived Mesenchymal stem cells (MSCs) in patient with lumbar intervertebral disc degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand and sign the consent form for this study
* Age :19-70, males and females
* Have chronic low back pain for at least 1 year
* Have failed 1 year of non-operative low back pain management
* Have degenerated intervertebral disc on T2-weighted MR images
* confirmed by positive discography
* Have significant lumbar instability at degenerated intervertebral disc

Exclusion Criteria:

* Have significant lumbar herniated intervertebral disc
* Women who are pregnant or breast feeding or planning to become pregnant during the study
* History or current evidence of alcohol or drug abuse or is a recreational user of illicit drugs or prescription medications
* Serious pre-existing medical conditions like Cardiovascular Diseases, Renal Diseases, Liver Diseases, Endocrine Diseases, Cancer and Diabetes Mellitus
* Participation in another clinical trial or treatment with a different investigational product within 30 days prior to inclusion in the study
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging | 24 weeks
  To evaluate the change of treated lumbar intervertebral discs using Magnetic Resonance Imaging (MRI) at 6 months post injection of MSCs.

SECONDARY OUTCOMES:
Changes of Neurological Functions | 24 weeks
  To evaluate the change of treated lumbar intervertebral discs using Muscle Test, Somatosensory Test, Deep Tendon Reflex and VAS (Visual Analogue Scale Score 0-10) at 6 months post injection of MSCs.
Safety evaluation | 24 weeks
  To determine the overall safety of Autologous Adipose Tissue Derived Mesenchymal Stem Cells carrier using physical examinations, vital signs, treatment emergent adverse events (TEAEs), and the results of clinical lab tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea